CLINICAL TRIAL: NCT07280494
Title: An Open-label, Clinical Study of CD7-targeted CAR-T Cells for the Treatment of Measurable Residual Disease of T-lymphoblastic Leukaemia/Lymphoma Post Allogeneic Stem Cell Transplantation
Brief Title: To Observe the CD7-targeted CAR-T Therapy in the Treatment of MRD Positive T-ALL/LBL Post Allo-HSCT
Acronym: S101MRD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Chief, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti CD7 CAR-T for MRD+ T-ALL
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: CD7+ T-ALL/LBL
Keywords: CD7; CAR T cell therapy; T-lymphoblastic leukemia/lymphoma; measurable residual disease; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Lymphoma; Neoplasm, Residual | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: A single group of patients receives a dose of 2e6 cells/kg NS CD7-targeted cell therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti CD7 CAR-T cells therapy (Experimental): eligible patients will be treated with CD7-targeted CAR-T cells
  Interventions: Drug: CAR-T Therapy

INTERVENTIONS:
Drug: CAR-T Therapy — autologous or donor-derived CD7-targeted CAR-T cells, single injection

SUMMARY:
To observe the efficacy and safety of CD7-targeted chimeric antigen receptor T cells in the treatment of T-lymphoblastic leukaemia/lymphoma with postive measurable residual disease positive post allogeneic stem cell transplantation

DETAILED DESCRIPTION:
This study will explore the efficacy and safety of a natural selection-targeted CD7 CART cell therapy for measurable residual disease after allogeneic hematopoietic stem cell transplantation in T-ALL/LBL. The dose of targeted CD7 CART cells is 2E6 cells/kg, with a single infusion.

ELIGIBILITY:
Inclusion Criteria:

* (1) The subject or the legal guardian understands and voluntarily signs the informed consent form (ICF).

  (2) Male or female, age ≥ 3 years at the time of signing the informed consent form.

  (3) Expected survival period of no less than 12 weeks. (4) ECOG performance score of 0-2 at the time of signing the ICF. (5) Confirmed as relapsed/refractory T-cell leukemia or lymphoma at the time of signing the ICF, meeting the following criteria:
  1. Bone marrow morphology examination at screening shows the proportion of primitive immature lymphocytes in the bone marrow < 5%, and positive for minimal residual disease of leukemia/lymphoma determined by flow cytometry.
  2. Tumor cells in the bone marrow or peripheral blood are CD7 positive as detected by flow cytometry.

     (6) Major organ functions must meet the following requirements:

  <!-- -->

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5× upper limit of normal (ULN).
  2. Total bilirubin ≤ 2× ULN.
  3. For adult subjects, the serum creatinine clearance rate ≥ 60 mL/min (Cockcroft-Gault formula) or serum creatinine ≤ 1.5× ULN; for children, the serum creatinine should be no more than 0.8 mg/dL for 2 to 6 years old, 1.0 mg/dL for 6 to 10 years old, 1.2 mg/dL for 10 to 13 years old, 1.5 mg/dL for 13 to 16 years old males, and 1.4 mg/dL for females over 13 years old; for males over 16 years old, it should be no more than 1.7 mg/dL.
  4. If the above organ function abnormalities are caused by infiltration of the primary disease, the decision on whether to include the subject in the study is made by the investigator.

     (7) Blood oxygen saturation > 92%. (8) Male subjects with reproductive capacity and female subjects of childbearing age must agree to use effective contraceptive measures from the time of signing the informed consent form until 2 years after the use of the study drug. Female subjects of childbearing age include premenopausal women and women within 2 years after menopause. The blood pregnancy test of female subjects of childbearing age at screening must be negative.

     Exclusion Criteria:
* Subjects with any of the following conditions will not be eligible for inclusion in this study.

  1. A history of CNS diseases, including but not limited to epilepsy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, and neuropathy. A history of diseases without related neurological symptoms before screening, such as lacunar infarction, etc., will be excluded at the discretion of the investigator.
  2. Any uncontrolled active infection within 4 weeks before signing the ICF or before apheresis.
  3. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at screening and peripheral blood hepatitis B virus (HBV) DNA above the detection limit, positive hepatitis C virus (HCV) antibody and positive HCV RNA, positive human immunodeficiency virus (HIV) antibody, cytomegalovirus (CMV) DNA above the detection limit, Epstein-Barr virus (EBV) DNA above the detection limit, and both specific and non-specific antibodies for Treponema pallidum positive need to be excluded.
  4. Clinically significant cardiovascular diseases, including any of the following:

     1. Corrected QTc interval ≥ 480 ms (QTc interval calculated by the Fridericia formula);
     2. New York Heart Association (NYHA) class II or higher heart failure;
     3. Unstable angina or acute myocardial infarction within 6 months before signing the ICF;
     4. Left ventricular ejection fraction (LVEF) < 50%;
     5. Uncontrolled hypertension (judged by the investigator based on the individual condition of the subject);
     6. Clinically significant or requiring antiarrhythmic treatment arrhythmias (such as sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes, and complete left bundle branch block, etc.).
  5. Allergy to any component of the drugs to be used in this study.
  6. Received any investigational drug treatment or other systemic anti-tumor treatment within 4 weeks before apheresis (or 5 half-lives of the drug, whichever is judged more appropriate by the investigator), except for bridging chemotherapy due to large tumor burden or rapid disease progression.
  7. Received extensive radiotherapy within 4 weeks before signing the ICF, except for local radiotherapy for symptom relief of non-target lesions during the study period.
  8. Received systemic corticosteroids (dose equivalent to or higher than 10 mg/day of prednisone) or other immunosuppressive drugs within 3 days before apheresis or during the study period, except for the following situations:

     1. Intranasal, inhaled, topical steroids or local steroid injections (such as intra-articular injections);
     2. Systemic corticosteroids at a dose not exceeding 10 mg/day of prednisone or its equivalent physiological dose;
     3. Steroids as prophylactic treatment for allergic reactions (such as pre-treatment before computed tomography [CT]);
     4. For the treatment of adverse reactions after reinfusion.
  9. Received major surgery within 4 weeks before signing the ICF (routine biopsy surgeries excluded), or expected to undergo major surgery during the study period.
  10. Had active tuberculosis infection within 1 year before signing the ICF (except for subjects with active tuberculosis infection more than 1 year ago and judged by the investigator to have no evidence of active tuberculosis at present).
  11. Received live attenuated vaccines within 4 weeks before signing the ICF or planned to receive live attenuated vaccines during the screening period.
  12. The investigator believes that the subject's complications or other conditions may affect compliance with the protocol or are not suitable for participation in this study.
  13. Pregnant or lactating.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
+1m MRD negtaive rate | 28 days post CAR-T infusion
  The MRD negative rate post CAR-T infusion

SECONDARY OUTCOMES:
+2m MRD negative rate | at 2 months post CAR-T infusion
  The MRD negative rate at 2 months post CAR-T infusion
+3m MRD negative rate | at 3 months post CAR-T infusion
  The MRD negative rate at 3 months post CAR-T infusion
survival | at 1 year post CAR-T infusion
  overall survival and progress free survival,non-relapse survival
relapse | at 1 year post CAR-T infusion
  the cumulative incidence of leukemia relapse
GVHD | 1 year post CAR-T infusion
  The incidence of grade III-IV acute GVHD and moderate to severe chronic GVHD.
hematological toxicity | 3 months post CAR-T therapy
  the incidenc and duration of Grade III-IV hematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided